CLINICAL TRIAL: NCT02775929
Title: An Open Label, Pilot Demonstration and Evaluation Project of Antiretroviral-based HIV-1 Prevention Among High-risk Serodiscordant African Couples
Brief Title: Partners Demonstration Project of PrEP and ART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); National Institute of Mental Health (NIMH) (NIH); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jared Baeten, Professor, Global Health, Medicine, & Epidemiology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001674; R01MH095507 (NIH)
Record Dates: First submitted 2016-05-10; First posted 2016-05-18 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: HIV Infection
Keywords: Tenofovir disoproxil; Emtricitabine; Pre-exposure Prophylaxis; Antiretroviral Therapy; HIV Prevention; FTC TDF; PrEP; HIV Infected Partners; HIV Uninfected Partners
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PrEP as a bridge to ART (Other): FTC-TDF PrEP for HIV uninfected partners and ART for HIV infected partners
  Interventions: Drug: FTC-TDF PrEP; Drug: ART

INTERVENTIONS:
Drug: FTC-TDF PrEP — FTC-TDF PrEP for HIV-1 uninfected partners
Drug: ART — ART for HIV-1 infected partners

SUMMARY:
The purpose of this protocol is to determine user preferences for antiretroviral therapy (ART) for HIV-1 infected partners and pre-exposure prophylaxis (PrEP) HIV-1 un-infected partners and to optimize targeted delivery and sustained use of these interventions.

DETAILED DESCRIPTION:
An open-label, prospective cohort study of higher-risk HIV-1 serodiscordant couples in order to determine barriers and facilitators to uptake and sustained adherence to ART for HIV-1 infected partners and daily oral PrEP for HIV-1 uninfected partners. The investigators developed a risk score tool to identify couples at highest risk for HIV-1 transmission. PrEP was offered as a 'bridge' to ART in the partnership - i.e., until ART initiation by the HIV-infected partner and for the first 6 months after ART is started; ART was recommended following national ART guidelines. A subset (up to 80 couples per site) was invited to participate in qualitative in-depth interview and focus group discussions.

ELIGIBILITY:
Inclusion Criteria:

For couples

* Risk score defining higher HIV-1 risk (≥6)
* Sexually active (defined as having had vaginal intercourse at least 6 times in the previous three months)
* Willing to enter the study as a couple and intending to remain as a couple for the next 12 months
* Did not participate in the Partners PrEP Study

For HIV-1 uninfected members of the couple (partner participants)

* Age ≥18
* Able and willing to provide written informed consent
* HIV-1 uninfected based on negative HIV-1 rapid tests, both at study screening and at the enrollment visit
* Adequate renal function, defined by normal creatinine levels and estimated creatinine clearance >60 mL/min
* Not infected with hepatitis B virus, as determined by a negative hepatitis B surface antigen test
* Not currently pregnant or breastfeeding
* Not currently enrolled in an HIV-1 prevention clinical trial
* Not currently using PrEP
* Enrollment of individuals with active and serious infections or active clinically significant medical problems will be at the discretion of the site investigator

For HIV-1 infected members of the couple (index participants)

* Age ≥18
* Able and willing to provide written informed consent
* HIV-1 infected based on positive rapid HIV-1 tests, according to national algorithm
* No history of WHO stage III or IV conditions
* Not currently using ART
* Not currently enrolled in an HIV-1 treatment study
* Note: current pregnancy and breastfeeding are permitted for HIV-1 infected partners

Exclusion Criteria:

* Otherwise not eligible based on the above inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1013 (Actual)
Dates: Start 2012-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Ability to recruit high-risk HIV-1 serodiscordant couples: Screen-to-eligible ratio. | 24 months
  High-risk couples defined by a validated risk scoring tool. Ability to recruit high-risk HIV-1 serodiscordant couples will be measured as screen-to-eligible ratio of HIV-1 serodiscordant couples.
Ability to recruit high-risk HIV-1 serodiscordant couples: Eligible couples who decide to enroll in the cohort. | 24 months
  High-risk couples defined by a validated risk scoring tool. We will measure the proportion of eligible couples who decide to enroll in the cohort.
Ability to recruit high-risk HIV-1 serodiscordant couples: Costs of screening and targeting high-risk couples decide to enroll in the cohort. | 24 months
  High-risk couples were defined by a validated risk scoring tool. The cost-effectiveness analysis will follow World Health Organization (WHO) guidelines and report summary estimates for the PrEP intervention which allow comparison to other strategies to decrease HIV-1 transmission among serodiscordant couples. Costs of offering and delivering PrEP as a bridging strategy to ART, including recruitment costs for targeting higher-risk couples and PrEP delivery and monitoring costs will be collected. The incremental cost-effectiveness ratio (ICER) per HIV related infection, death and Disability-Adjusted Life Year (DALY) averted will be estimated. Results will be reported as the ICER of PrEP compared to current practice per incident HIV-1 case, HIV related death and DALY averted.
User preferences for ART initiation for HIV-1 infected partners and PrEP for HIV-1 uninfected partners: preferred ART-based HIV prevention method. | 24 months
  Measure the number of couples choosing to use PrEP or ART for HIV-1 prevention or both.
User preferences for ART initiation for HIV-1 infected partners and PrEP for HIV-1 uninfected partners: reasons for choice and concerns about both methods. | 24 months
  Quantitative questionnaire will be used to elicit reasons for the choice and concerns about both methods. Reasons for or concerns about both methods measured as proportion of participants reporting a particular reason for or concerns about both methods
PrEP initiation by HIV uninfected partners. | 24 months
  Measure the number of HIV-1 uninfected partners initiating PrEP.
  Proportion of samples with detectable and quantifiable PrEP levels
PrEP adherence: Self-reported missed doses of PrEP. | 24 months
  Measure the proportion of visits when HIV-uninfected partner reported missing 1) any dose of PrEP in the prior quarter 2) 2 or more consecutive doses of PrEP.
PrEP adherence: Detectable and quantifiable PrEP levels in plasma. | 24 months
  Measure the proportion of plasma samples of HIV-1 uninfected partners with detectable and quantifiable PrEP levels.
PrEP adherence: PrEP hold. | 24 months
  Measure the total number of HIV-1 uninfected partners with PrEP hold designated as a safety issue.
ART initiation. | 24 months
  Measure the number of HIV-1 infected partners initiating ART.
ART Adherence. | 24 months
  Measure the number of HIV-1 infected partners with suppressed plasma HIV-1 RNA levels.
Correlates of preferences, uptake and adherence to ART and PrEP: Sexual frequency. | 24 months
  Proportion of visits when participants report having sex.
Correlates of preferences, uptake and adherence to ART and PrEP: Condom use frequency. | 24 months
  Proportion of visits when participants report having condomless sex.
Correlates of preferences, uptake and adherence to ART and PrEP: Outside partners for HIV-1 uninfected partners. | 24 months
  Proportion of visits when HIV-1 uninfected partners report outside partners.
Correlates of preferences, uptake and adherence to ART and PrEP: Gender of the HIV-1 uninfected partner. | 24 months
  Proportion of couples in which the HIV-1 uninfected partner is female.
Correlates of preferences, uptake and adherence to ART and PrEP: Fertility intentions. | 24 months
  Proportion of couples with desire to conceive a child.
Correlates of preferences, uptake and adherence to ART and PrEP: Relationship dissolution. | 24 months
  Number of couples continuing their relationship during follow up.
Correlates of preferences, uptake, and adherence to ART and PrEP: Depression and substance use. | 24 months
  Annual interviewer-administered questionnaire to collect depression and substance use indicators. Measure proportion of participants with depression and substance use.
Correlates of preferences, uptake and adherence to ART and PrEP: ART initiation by HIV-1 infected partner. | 24 months
  Proportion of HIV-1 infected partners initiating ART.
Correlates of preferences, uptake and adherence to ART and PrEP: Number of children. | 24 months
  Proportion of partnership reporting to have children at baseline.
Correlates of preferences, uptake and adherence to ART and PrEP: CD4 count. | 24 months
  Proportion of HIV infected partners with CD4 count >200, >350, >500.
Correlates of preferences, uptake and adherence to ART and PrEP: WHO stage of HIV-1 infected partner. | 24 months
  Proportion HIV-1 infected partners with WHO HIV-1 stage 1, 2, 3, or 4.
Feasibility to PrEP discontinuation in couples when the HIV-1 infected partner initiates ART. | 24 months
  We will conduct in-depth interviews and focus group discussions. Qualitative analyses will identify and describe key themes and explore variation within themes of participants' attitudes and understanding of PrEP discontinuation.
PrEP use and pregnancy: HIV-1 infection. | 24 months
  Number of HIV-1 infections among women who continue PrEP in pregnancy.
PrEP use and pregnancy: Congenital abnormalities among infants born to female Participants taking PrEP. | 24 months
  Infant outcomes measured as the number of live-born infants born to female participants taking PrEP that had any congenital anomalie.
PrEP use and pregnancy: Any serious adverse event. | 24 months
  Number of women who continue PrEP in pregnancy with any serious adverse event.
Infant growth for women who continue PrEP in pregnancy: Length. | 24 months
  Length of infants born to female Participants taking PrEP. The slope of the linear model of the growth of infants (length) during the entirety of follow-up. The length of the infant measured as a z-score, in terms of standard deviations from the age and gender specific median using the World Health Organization growth curve, accounting for skewness. The slope, representing the change over time of the z-score, will be calculated using all available z-scores over study duration and regressing against study month.
Infant growth for women who continue PrEP in pregnancy: Weight. | 24 months
  The slope of the linear model of the growth of infants (weight) during the entirety of follow-up. The weight of the infant was measured as a z-score, in terms of standard deviations from the age and gender specific median using the World Health Organization growth curve, accounting for skewness. The slope, representing the change over time of the z-score, will be calculated using all available z-scores over study duration and regressing against study month.
Infant growth for women who continue PrEP in pregnancy: Head circumference. | 24 months
  The slope of the linear model of the growth of infants (head circumference) during the entirety of follow-up. The head circumference of the infant will be measured as a z-score, in terms of standard deviations from the age and gender specific median using the World Health Organization growth curve, accounting for skewness. The slope, representing the change over time of the z-score, will be calculated using all available z-scores over study duration and regressing against study month.

CONTACTS AND LOCATIONS:
Overall Officials: Jared M Baeten, MD, PhD, Principal Investigator — University of Washington
Locations (4):
- Kenya (2):
  - Kemri-Ucsf, Kisumu
  - Partners in Prevention-Thika, Thika
- Uganda (2):
  - Kabwohe Clinical Research Center, Bushenyi
  - Partners in Prevention-Infectious Diseases Institute LTD, Kampala

IPD SHARING:
Plan to Share IPD: Yes
Data from the Partners Demonstration Project are available by contacting the International Clinical Research Center at the University of Washington (icrc@uw.edu).

REFERENCES:
- [Derived] Nakku-Joloba E, Pisarski EE, Wyatt MA, Muwonge TR, Asiimwe S, Celum CL, Baeten JM, Katabira ET, Ware NC. Beyond HIV prevention: everyday life priorities and demand for PrEP among Ugandan HIV serodiscordant couples. J Int AIDS Soc. 2019 Jan;22(1):e25225. doi: 10.1002/jia2.25225. PMID 30657642